CLINICAL TRIAL: NCT02375906
Title: Hepatitis Delta Registry and Research Network- Observational Study
Brief Title: The Hepatitis Delta International Network
Acronym: HDIN
Status: Completed | Type: Observational
Sponsor: HepNet Study House, German Liverfoundation (Network)
Collaborators: German Center for Infection Research (Other); Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: HepNet-HDIN
Record Dates: First submitted 2015-02-19; First posted 2015-03-03 (Estimated); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: Hepatitis D
Keywords: HDV, hepatitis delta
MeSH Terms: conditions — Hepatitis D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Hepatitis delta is a major health problem, not only because of the severity of the disease, but also due to the lack of effective antiviral treatment. To improve the current therapeutic options, a better understanding of the pathophysiology is essential. Reliable research in this direction is only possible with large patient study groups. However, given the geographic distribution of hepatitis delta, larger patient cohorts would only be possible through multicenter collaboration.

DETAILED DESCRIPTION:
The hepatitis international network cohort is a multicenter, observational study that will build up a research registry of HDV patients all over the world.

The aims of this project are:

i. Collect clinical information from hepatitis delta patients from multiple centers distributed worldwide in order to build up a large database that will enable and facilitate further research on chronic hepatitis delta.

ii. To better inform patients about their viral infection, present status and evolution of liver disease throughout time. To give them the tools needed to inform other peers and medical professionals about the significance and consequences of a chronic hepatitis delta infection.

iii. To allow the participating physicians to track course of the disease, therapies, signs and symptoms of the hepatitis delta patients included by their center.

ELIGIBILITY:
Inclusion Criteria:

• Positive HBs antigen and antiHDV for longer than 6 months.

Exclusion Criteria:

Absence of any cause of relevant liver disease other than HDV (i.e. hemochromatosis, autoimmune hepatitis, alcoholic or toxic liver disease, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic hepatitis delta will be screened regardless of HDV or HBV genotype
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Proportion of chronic hepatitis B patients with chronic hepatitis D infection worldwide | 10 years

SECONDARY OUTCOMES:
HDV-RNA HBsAg | 10 years
HBV-DNA | 10 years
Proportion of treated chronic hepatitis B patients with chronic hepatitis D infection worldwide | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Manns, Prof. Dr., Principal Investigator — Hannover Medical School
Locations (18):
- Medical University of Vienna; Internal Med.III, Vienna, Austria
- Antwerpen University Hospital, Edegem, Belgium
- Centro de Pesquisa em Medicina Tropical, Rondônia, Brazil
- Medical Center Mrcheveli, Tbilisi, Georgia
- Germany (4):
  - Medizinisches Infektiologiezentrum, Berlin
  - Medizinische Klinik I Charite- Campus Benjamin Franklin, Berlin
  - Universitätsklinikum Giessen-Marburg, Giessen
  - Medizinische Hochschule Hannover, Hanover
- Dep.of Medicine University of Thessalony, Larissa, Greece
- Italy (3):
  - Centro di ricerca per lo studio della Epatiti, Bologna
  - Gastroenterology Casa Sollievo della Sofferenza Hospital, San Giovanni Rotondo
  - A.O.U. Citta della Salute e della Scienza di Torino, Torino
- The University of Medicine "Nicolae Testimitanu", Chisinau, Moldova
- Pakistan (2):
  - Dept.of Medicine Aga Khan University, Karachi
  - Liverstomach Clinic, Karachi
- Clinical Hospital of Infectious Disease "dr. Victor Babes", Bucharest, Romania
- Hospital Vall d´Hebron, Barcelona, Spain
- Vietnamese-German Center for Medical Research, Hanoi, Vietnam

REFERENCES:
- [Result] Wranke A, Pinheiro Borzacov LM, Parana R, Lobato C, Hamid S, Ceausu E, Dalekos GN, Rizzetto M, Turcanu A, Niro GA, Lubna F, Abbas M, Ingiliz P, Buti M, Ferenci P, Vanwolleghem T, Hayden T, Dashdorj N, Motoc A, Cornberg M, Abbas Z, Yurdaydin C, Manns MP, Wedemeyer H, Hardtke S; Hepatitis Delta International Network. Clinical and virological heterogeneity of hepatitis delta in different regions world-wide: The Hepatitis Delta International Network (HDIN). Liver Int. 2018 May;38(5):842-850. doi: 10.1111/liv.13604. Epub 2017 Oct 26. PMID 28963781